CLINICAL TRIAL: NCT06201260
Title: Effects of Intermittent Pneumatic Compression Following Exercise-induced Muscle Damaged
Acronym: IPC4sports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDFM_003; IPC (Other: University of Maia)
Record Dates: First submitted 2023-11-24; First posted 2024-01-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC (Experimental): a 30 min high-pressure IPC protocol
  Interventions: Other: intermittent pneumatic compression protocol
- placebo (Placebo Comparator): A 30 min placebo
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: intermittent pneumatic compression protocol — A 30 min IPC protocol at about 200mmHg
  Arms: IPC
Other: Placebo treatment — The electrodes of an electrostimulation device (SP 4.0, Compex, Guildford, United Kingdom) will be positioned on participants' quadriceps. Participants will be informed that they are engaging an innovative microcurrent treatment. This procedure will last for 30 min.
  Arms: placebo

SUMMARY:
This study aims to assess the recovery kinetics following an exercise-induced muscle damage activity (using flywheel) on active healthy university students.

The main questions are:

- Is intermittent pneumatic compression superior to a placebo recovering from EIMD? Participants will perform a fatiguing protocol using flywheel and recover with either intermittent pneumatic compression or with a placebo treatment (micro-current treatment, but the device turned off). They will perform several performance tests before, following the recovery period, and at the 24h and 48h following the intervention

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participating in this study, participants should not have been recently injured, and should engage physical activity regularly (>3 times/week).

Exclusion Criteria:

* Inactive participants
* Younger than 18 years old or older than 27 years old

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male gender
Enrollment: 33 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction (knee extension) | 10 minutes before the fatigue protocol, following the recovery protocol (30 minutes post), 24 hours and 48 hours post intervention
  Measures of isometric strength
Countermovement jump | 10 minutes before the fatigue protocol, following the recovery protocol (30 minutes post), 24 hours and 48 hours post intervention
  Jump height
Broad Jump | 10 minutes before the fatigue protocol, following the recovery protocol (30 minutes post), 24 hours and 48 hours post intervention
  Horizontal jump
Soreness scale | 10 minutes before the fatigue protocol, following the recovery protocol (30 minutes post), 24 hours and 48 hours post intervention
  Likert scale of muscle soreness - the scale ranges from from 0 (a complete absence of soreness) to 6 (a severe pain that limits the ability to move)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Portugal